CLINICAL TRIAL: NCT02217553
Title: The Effect of Vitamin D Supplementation on HIV-associated Platelet Hyperreactivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Mohammad Ghozali, Medical Doctor, Universitas Padjadjaran
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1402001
Record Dates: First submitted 2014-08-12; First posted 2014-08-15 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Blood Platelet Disorders; Vitamin D Deficiency
Keywords: platelet; P-selectin; platelet-fibrinogen binding; platelet-monocye aggregate formation; vitamin D
MeSH Terms: conditions — Blood Platelet Disorders; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- vitamin D (cholecalciferol) (Experimental): All study participants will receive vitamin D supplementation (soft gel capsule containing cholecalciferol 400 IU) to be consumed 2 soft gel capsules daily for three consecutive months. The effect on the platelet parameters specified above will be determined before start cholecalciferol supplementation and after three months.
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — The study participants will receive 180 soft gel cholecalciferol capsules, to be taken 2 capsules once a day for 90 days
  Other Names: Teorol

SUMMARY:
Platelets play pivotal role in atherosclerosis and acute cardiovascular events. Platelet hyperreactivity and increase platelet-monocyte aggregate (PMA) formation are found in HIV infected patients, which may contribute to the excess cardiovascular risk. Low level of vitamin D has been associated with the presence of cardiovascular diseases. The aim of our study is to determine the effect of vitamin D supplementation on platelet activation, platelet reactivity and platelet-leukocyte complex formation in asymptomatic HIV-infected patients treated with ART

DETAILED DESCRIPTION:
1. Study design A prospective intervention study. HIV-infected patients using ART and who come for follow-up at the Teratai HIV clinic will be asked to participate in the study. All study participants will receive vitamin D supplementation (soft gel capsule containing cholecalciferol 400 IU) to be consumed 2 soft gel capsules daily for three consecutive months. The effect on the platelet parameters specified above will be determined before start cholecalciferol supplementation and after three months.
2. Duration of study Usually, 150 HIV-infected patients are treated with ART every week at the Teratai HIV clinic of the Hasan Sadikin Hospital Bandung Indonesia. Between half January 2014 and end of February 2014, 50 patients will be enrolled in this study. We hypothesize that this period is long enough to include 50 patients for the present study. Supplementation will take place between March and May and analysis will be done in June and July. A summary of duration of study is depicted in the study timeline.
3. Study population The study population consists of adult HIV-infected patients treated with ART enrolled at HIV polyclinic at Hasan Sadikin General Hospital, Bandung, Indonesia.
4. Sample size calculation Our sample size calculation is based on the primary outcome, which is the area under the curve (AUC) of the platelet reactivity curve with P-selectin (CD62P) as platelet activation marker and ADP as platelet agonist. In a cohort of Dutch HIV-infected patients we found a mean AUC of 2500 with an SD of 660. Assuming that a decrease in AUC of 2500 to 2100 upon supplementation of vitamin D is clinically relevant, a sample size of 23 would be sufficient using a paired design with α 0.05 and a power of 80%.
5. Methods Study parameters/endpoints

   There are two study parameters applied in this study:
   1. Platelet reactivity, expressed as the membrane expression of the platelet activation markers CD62P (P-selectin) and fibrinogen binding to integrin αIIbβ3, to stimulation with increasing concentration of platelet agonists ADP.
   2. Platelet-monocyte complexes.
6. Study procedures

   a. Enrolment of patients During a scheduled routine polyclinic visit, the treating internist will identify patients fulfilling inclusion criteria. He/she will explain the background and objectives of the study to the patient. In case patients opt to participate, the patient will then be asked to read and undersign the informed consent form.

   Venous blood (three tubes of 3 mL each) will then drawn for study purpose at enrolment and after three months supplementation for:
   1. 25-hydroxyvitamin D level (3 ml serum)
   2. Platelet assays as specified above (3 ml CTAD)
   3. Full blood count and CD4 cells (3 ml EDTA) In many instances, this will not require an extra venepuncture as blood is usually collected for planned blood analysis for routine clinical care during regular polyclinic visits.

   Measurements and analysis consist of 25-hydroxyvitamin D level, platelet reactivity, and platelet-monocyte complexes will be done when the patients participate in the study. The study participants will receive 180 soft gel cholecalciferol capsules, to be taken 2 capsules once a day for 90 days as stated above.

   As stated above, the second blood analysis will take place three months later after vitamin D supplementation is completed.

   b. Collection of blood samples for vitamin D level analysis As much as 3mL additional blood is withdrawn while applying venepuncture for routine CD4+ measurement. Collected blood is stored using red top serum tube without anticoagulant. This will take place at enrolment (day 0) and after 3 months vitamin D supplementation. Each day of blood withdrawal, the collected tubes are stored temporarily in wet-iced box prior transfer to laboratory for vitamin D analysis. At the end of the policlinic day, all tubes are transferred to the laboratory for serum separation. Then, separated serum is stored so 25-hydroxyvitamin D measurements can be done later. All samples are analysed for 25-hydroxyvitamin D measurements as well as other vitamin D metabolites such as free 25-hydroxyvitamin D measurements. Such analysis can not be done in Indonesia and therefore samples will be shipped to the Netherlands for this purpose.

   c. Collection of blood samples for platelet function analysis As specified under study parameters above, platelet function analysis can be performed from one 3mL citrate-anticoagulated blood tube. This will take place at enrolment (day 0) and after 3 months vitamin D supplementation. Each withdrawn blood from the patient, the tube is directly transferred to the laboratory for platelet function within 30 minutes.

   d. Full blood count and CD4 cell measurements These measurements are part of routine care and will be done in the routine haematological laboratory using 3 ml EDTA blood.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* Treated with suppressive first-line ART for at least 12 months
* Compliant to ART and procedures of Teratai clinic
* No signs or symptoms

Exclusion Criteria:

* Use of aspirin or other platelet function inhibitors.
* Any sign or symptom
* Known active opportunistic infection
* Active illicit drug users or any other comorbidity
* History of failing ART or non-compliance.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-12; Primary Completion 2014-02 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The effect of vitamin D supplementation on HIV-associated platelet hyperreactivity | Three months
  Mean Fluorescence Intensity of the platelet reactivity curve before and after receiving vitamin D

SECONDARY OUTCOMES:
The effect of vitamin D supplementation in platelet-monocyte aggregate formation | three months
  Mean fluorescence intensity of platelet-monocyte aggregate before and after vitamin D supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Andre van der Ven, Professor, Study Chair — Radboud University Medical Center; Quirijn de Mast, Doctor, Study Director — Radboud University Medical Center; Rudi Wisaksana, Doctor, Study Director — Universitas Padjadjaran; Agnes R Indrati, Doctor, Study Director — Universitas Padjadjaran
Locations (1):
- Klinik Teratai Hasan Sadikin General, Bandung, West Java, Indonesia

REFERENCES:
- See also: Official web site of Faculty of Medicine, Universitas Padjadjaran — http://www.fk.unpad.ac.id
- See also: Official web site of Radboud University Medical Center — http://www.radboudumc.nl